CLINICAL TRIAL: NCT03008928
Title: The Efficacy of the Alcooquizz App to Reduce Hazardous Alcohol Consumption: Randomized Controlled Trial
Brief Title: The Efficacy of the Alcooquizz App to Reduce Hazardous Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 108/2016
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention
- Alcooquizz app (Experimental): Alcooquizz is a smartphone app designed to promote reductions in alcohol consumption among people who drink in a hazarzdous fashion
  Interventions: Behavioral: Alcooquizz

INTERVENTIONS:
Behavioral: Alcooquizz
  Arms: Alcooquizz app

SUMMARY:
New technologies offer potential ways to provide and deliver preventative interventions. With respect to unhealthy alcohol use, offering people tools to assess and manage their risk at any given time using their smartphone may represent an additional opportunity to disseminate preventative interventions. Nevertheless, there is a lack of knowledge on the acceptability and efficacy of smartphone applications for unhealthy alcohol use. Alcooquizz, a smartphone app, has been previously evaluated using a before/after design without randomization, with participants reporting reductions in drinking over time. The current trial proposes to conduct an RCT, comparing reductions in alcohol consumption between participants provided access to Alcooquizz to a no intervention control.

Participants will be recruited through Amazon's MTurk crowdsourcing platform. Potential participants identified as problem drinkers based on an initial survey will be invited to complete another survey in 6 months time. Those who agree to be followed-up will be randomized to be provided a link to download the Alcooquizz app or to a no link control condition. At six-months post-baseline, the MTurk portal will be used to send invitation emails that contain a link to the follow-up survey that asks about their drinking and their impressions of the app. The primary hypothesis to be tested is that participants receiving access to the Alcooquizz app will report a greater level of reduction in number of drinks in a typical week between the baseline survey and six-month follow-up as compared to participants in the no information control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Typically consumes 15 or more drinks per week,
* Willingness to complete a 6-month follow-up survey

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in number of drinks in a typical week from baseline | 6 months
  Sum of number of drinks consumed in a typical week

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schell C, Godinho A, Cunningham JA. To thine own self, be true: Examining change in self-reported alcohol measures over time as related to socially desirable responding bias among people with unhealthy alcohol use. Subst Abus. 2021;42(1):87-93. doi: 10.1080/08897077.2019.1697998. Epub 2020 Feb 10. PMID 32040383